CLINICAL TRIAL: NCT02996708
Title: Assessment of the Benefit of Teleconsultations for Children With Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: TLM Prometted
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Autism Spectrum Disorder; Child Autism
Keywords: Telemedicine; Health economics
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group with teleconsultation - before period
- Group without teleconsultation - before period
- Group with teleconsultation - after period
- Group without teleconsultation - after period

SUMMARY:
The purpose of this study is to determine whether Teleconsultation would a)be effective and cost-effective by increasing the proportion of patients with Autism Spectrum Disorders having a correct follow-up, and less transportation, and b) get a high satisfaction from the parents and from the professionals

ELIGIBILITY:
Inclusion Criteria:

* All residents of medico-social structures accepting children and adolescent with autism disorders

Exclusion Criteria:

* Refusal of parents that their child use telemedicine
* Refusal of parents that their child participate to the research

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Residents of medico-social structure accepting children and adolescent with autism disorders
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite score: CARS, VABS evaluated once a year and ADI-R at least once in the lifetime | One year after the start of the "before" period and one year after the start of the "after" period
  Score equals 1 if all three evaluations are performed, 0 otherwise

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Doyen, MD, Principal Investigator — Hôpital Sainte Anne
Locations (6):
- France (6):
  - IME notre Ecole, Carrières-sous-Poissy
  - Association Agir et Vivre l'Autisme, Chambourcy
  - IME Eclair, Collégien
  - Association UNI-TEDS, Dammarie-les-Lys
  - Hôpital Sainte Anne, Paris
  - IME Le Reverdi, Vert-Saint-Denis

IPD SHARING:
Plan to Share IPD: No